CLINICAL TRIAL: NCT04264832
Title: Department of Traditional Chinese Medicine (TCM), Center for Reproductive Medicine, Department of Obstetrics and Gynaecology, Peking University Third Hospital, Beijing 100191, China.
Brief Title: Body Fat Distribution and Its Associated Factors in Chinese Women With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Peking TCM
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-03

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: fat distribution; insulin resistance; negative emotion; polycystic ovary syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: Participants were eligible if they met the Rotterdam diagnostic criteria of polycystic ovary syndrome (PCOS) and meet the inclusion and exclusion criteria , and all study participants received questionnaires and underwent the physical, transvaginal ultrasound and body composition examination. Blood samples were collected for analysis of metabolic markers, metabonomics and hormones.
  Interventions: Other: Clinical data collection
- control group: The control group participants are normal women and had no history of any type of diabetes, cardiovascular disease (myocardial infarction, unstable angina, stroke or cardiovascular revascularization), stage 2 hypertension , malignant disease or severe renal or hepatic disease. They accepted the same examinations as the observation group.
  Interventions: Other: Clinical data collection

INTERVENTIONS:
Other: Clinical data collection — Basic characteristics: Participants were carefully characterized with regard to a general health history, a medical history, clinical, demographic and anthropomorphic measurements, skin problems (hirsutism is modified by Ferriman-Gallwey (mF-G) score , global acne score and premature alopecia).
  A transvaginal ultrasound scan was performed on every participant during a clinical examination to determine the number of follicles and ovarian volume.
  Metabolic and other assessments: General gynecological examination, prolactin, thyroid, androgen, LH, FSH, DA, 5-HT, metabonomics, glucose, insulin, triglyceride (TG), LDL and HDL were determined, OGTT was performed.
  Questionnaires: The perceived stress scale(Chinese 14-item PSS), self-rating anxiety scale (SAS）, self-rating depressive scale(SDS) were used to assess the participants' mental health status. The MOS item short from health survey (SF-36) was used to assess the quality of life .

SUMMARY:
To investigate the body fat distribution in chinese women with polycystic ovary syndrome (PCOS) and the association of those distribution with metabolic parameters, microeconomics, hormone profiles and psychological state.

DETAILED DESCRIPTION:
The polycystic ovary syndrome (PCOS) is one of the most common endocrine and metabolic disorders in women of reproductive age. It is also one of the leading causes of anovulatory infertility and secondary amenorrhea, which represent major stress factors in the female life. In the previous studies, the investigators found that PCOS patients showed decreased quality-of-life and increased psychological disturbances compared with healthy controls. Body mass index (BMI) was associated with emotional disorders and physical aspects of quality-of-life and negative emotions were negatively correlated with BMI in PCOS patients.These results prompted that PCOS could be separated into at least two subtypes by the fat content. So the investigators expand the epidemiological investigation for comparing the body composition between the PCOS and the normal women, and finding specific biological indicators in different subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years
* For the PCOS group, PCOS diagnosis according to Rotterdam criteria 2003 with at least two of the following three symptoms: (1) infrequent ovulation or anovulation; (2) hyperandrogenism or clinical manifestations of high blood androgen; (3) ultrasound findings of polycystic ovaries in 1 or 2 ovaries, or ≥12 follicles measuring 2 to 9 mm in diameter, and/or ovarian volume ≥10 mL

Exclusion Criteria:

* Exclusion of other endocrine disorders such as androgen secreting tumors, suspected Cushing's syndrome and non-classic congenital adrenal hyperplasia (17-hydroxyprogesterone < 3nmol/L) thyroid dysfunction and hyperprolactinemia.
* Type I diabetes or not well controlled type II diabetes
* Stage 2 hypertension (resting blood pressure ≥160/100mmHg)
* Psychiatric diagnoses or using psychiatric medications including antidepressants
* Pharmacological treatment (cortizone, antidepressant, other antidiabetic treatment such as insulin and acarbose, hormonal contraceptives, hormonal ovulation induction or other drugs judged by discretion of investigator) within 12 weeks. Depo Provera or similar within 6 months.

The control group are non- PCOS normal women (age 18-45) and meet the same exclusion criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: a cross-sectional study was conducted in women of reproductive age (19- 45 years) from the Peking university third hospital
Sampling Method: Non-Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
body fat content and ratio | Baseline
  Examined with a body composition analyzer (Tanita Corporation, model MC-180, Japan)

SECONDARY OUTCOMES:
Body mass index (BMI) | Baseline
  Weight in kilograms divided by the square of height in meters, reported in kg/m2
Waist circumference(WC) | Baseline
  Waist circumference（WC）reported in cm, refers to the horizontal circumference along the midpoint of the connection line of the anterior superior iliac crest through the lower costal margin of the calm breathing state when standing. Recumbent position is the abdominal circumference through the girth of the navel.
Hip circumference | Baseline
  Hip circumference reported in cm, and when measured, the legs are upright and closed together, the arms are naturally pendulous, and the tape measure is placed horizontally on the pubic symphysis in front and the gluteus maximus in the back.
Waist-hip ratio (WHR) | Baseline
  Waist-to-hip ratio
Fat content and ratio of trunk | Baseline
  Examined with a body composition analyzer (Tanita Corporation, model MC-180, Japan)
Follicle stimulating hormone (FSH) | Baseline
  Examined with the blood sample
luteinizing hormone (LH) | Baseline
  Examined with the blood sample
Progestin (P) | Baseline
  Examined with the blood sample
Estrogen (E2) | Baseline
  Examined with the blood sample
Prolactin (PRL) | Baseline
  Examined with the blood sample
Androgen(T) | Baseline
  Examined with the blood sample
Androstenedione (A2) | Baseline
  Examined with the blood sample
Glucose | Baseline
  Examined with the blood sample
Insulin | Baseline
  Examined with the blood sample
HOMA-IR | Baseline
  calculation of HOMA-IR: [fasting insulin (μU/mL) × fasting glucose (mmol/L)] / 22.5)
HOMA- β | Baseline
  calculation of HOMA-β: 20 × fasting insulin (mU/mL) / (fasting plasma glucose (mmol/L) - 3.5) (%)
total cholesterol | Baseline
  examined with the blood sample
triglycerides | Baseline
  examined with the blood sample
high density lipoprotein (HDL) | Baseline
  examined with the blood sample
low density lipoprotein (LDL) | Baseline
  examined with the blood sample examined with the blood sample
β-endorphin | Baseline
  examined with the blood sample
5- hydroxytryptamine (5-HT) | Baseline
  examined with the blood sample
Dopamine(DA) | Baseline
  examined with the blood sample
lipometabonomics | Baseline
  examined with the blood sample
bile acid | Baseline
  examined with the blood sample (fasting plasma glucose (mmol/L) - 3.5) (%)
FerrimanGallwey (FG )value | Baseline
  To determine changes in women's hairy with FG rating scale (0-36 score), the higher, the worse
short form-36 (SF36) | Baseline
  determine the health quality of life by the questionnaire of SF36 (0-100 score), the higher, the better
Self-Rating Anxiety Scale (SAS) | Baseline
  determine the anxiety level with the questionnaire of SAS (20-100 score), the higher, the worse.
Self-Rating Depress Scale (SDS) | Baseline
  determine the depress level with the questionnaire of SDS (20-100 score), the higher, the worse
Preserved Stress Scale (PSS) | Baseline
  determine the stress level with the questionnaire of SDS (14-56 score), the higher, the worse

CONTACTS AND LOCATIONS:
Overall Officials: Haolin Zhang, Study Director — Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided whether to share the data

REFERENCES:
- [Derived] Yang S, Zhang H, Shi L, Yang Y, Lu Y, Qiu W, Fukuzawa I, Zhou L, Xin X, Ding N, Luo L, Wang W, Zhang H. Menstrual disorder is associated with blood type in PCOS patients: evidence from a cross-sectional survey. BMC Endocr Disord. 2025 Mar 24;25(1):77. doi: 10.1186/s12902-025-01898-0. PMID 40122801
- [Derived] Zhang H, Qiu W, Zhou P, Shi L, Chen Z, Yang Y, Lu Y, Zhou L, Zhang H, Cheng M, Ye Y, Li R. Obesity is associated with SHBG levels rather than blood lipid profiles in PCOS patients with insulin resistance. BMC Endocr Disord. 2024 Nov 25;24(1):254. doi: 10.1186/s12902-024-01789-w. PMID 39587600
- [Derived] Zhang H, Wang W, Zhao J, Jiao P, Zeng L, Zhang H, Zhao Y, Shi L, Hu H, Luo L, Fukuzawa I, Li D, Li R, Qiao J. Relationship between body composition, insulin resistance, and hormonal profiles in women with polycystic ovary syndrome. Front Endocrinol (Lausanne). 2023 Jan 9;13:1085656. doi: 10.3389/fendo.2022.1085656. eCollection 2022. PMID 36699018